CLINICAL TRIAL: NCT06122792
Title: Preemptive Transjugular Intrahepatic Portosystemic Shunt for Gastric Variceal Bleeding in Patients With Cirrhosis: A Multicenter Randomized Trial
Brief Title: Preemptive TIPS for Gastric Variceal Bleeding in Patients With Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: Beijing YouAn Hospital (Other); Renmin Hospital of Wuhan University (Other); Second Affiliated Hospital of Nanchang University (Other); Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pTIPS-GV
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Portal Hypertension; Gastric Varices Bleeding; Portosystemic Shunt
MeSH Terms: conditions — Hypertension, Portal | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (Active Comparator): Standard treatment to achieve initial hemostasis: vasoactive drugs (somatostatin or terlipressin) + endoscopic hemostasis according to the center protocol.
  Standard combined endoscopic and pharmacological therapy as secondary prophylaxis (carvedilol + repeated endoscopic injection of tissue adhesives until the eradication of the gastric varices).
  Interventions: Procedure: standard second prophylaxis
- Preemptive TIPS (Experimental): Standard treatment to achieve initial hemostasis: vasoactive drugs (somatostatin or terlipressin) + endoscopic hemostasis according to the center protocol.
  Performance of TIPS in the first 72 hours following initial endoscopic hemostasis.
  Interventions: Procedure: preemptive TIPS

INTERVENTIONS:
Procedure: preemptive TIPS — The TIPS procedure should be performed within 72 hours after the initial endoscopic examination or treatment. An 8 mm Viatorr stent will be used for TIPS establishment. The aim will be to reduce the portal pressure gradient below 12 mm Hg. Embolization, either with coils or glue, can be performed, if it is felt necessary, especially in patients where portography shows the filling of large portosystemic collaterals feeding the varices. After TIPS, anticoagulation will not be used as a rule but is allowed if the attending physician thinks that it is warranted.
  Other Names: early TIPS
  Arms: Preemptive TIPS
Procedure: standard second prophylaxis — Patients will receive vasoactive drugs up to 5 days; then a non-selective beta-blocker (carvedilol) will be started with an initial dose of 6.25 mg, the dose of propranolol will be increased to 12.5 mg.
  The second elective session of endoscopic injection of tissue adhesives will be performed within the first 28 days after the initial endoscopic treatment. The following sessions will be performed at 28 +/- 3 days intervals until variceal eradication. Once eradication is achieved, endoscopic monitoring will be performed every 6 months. If varices reappear, new endoscopic injection of tissue adhesives will be performed.
  Other Names: endoscopy plus drug treatment
  Arms: Standard Therapy

SUMMARY:
The prevalence of gastric varices is approximately 20%. It is important to note that gastric varices tend to bleed more severely, have a higher morbidity and mortality rate, and have a 35% to 90% risk of rebleeding after the cessation of acute hemorrhage. Because of the relatively low prevalence of gastric varices, the existing clinical studies have many deficiencies, and there is much controversy in the academic community, the optimal treatment and prevention strategies for gastric varices have not yet been fully defined.

In the last few years, important advances have been made in the treatment and prevention of gastric variceal bleeding in patients with cirrhosis. Experts agree that the combination of pharmacological and endoscopic injection of tissue adhesives should be the first line of therapy in the acute bleeding episode from isolated gastric varices (IGV1) or type 2 gastroesophageal varices (GOV2) varices; whereas transjugular intrahepatic portosystemic shunt (TIPS) is considered a rescue therapy. TIPS has been shown to effectively prevent variceal rebleeding but with a potential increase in the incidence of hepatic encephalopathy and/or liver failure. In this sense, a recent randomized controlled trial (RCT) in fundal variceal bleeding showed that an early TIPS, performed during the first 5 days after patient admission resulted in a significant decrease in failure to control bleeding and early and late rebleeding. However, the study was conducted for 4 years and only included 25 patients. Due to insufficient sample size, it was unable to reflect whether priority TIPS can bring survival benefits to patients with gastric variceal bleeding. Therefore, there is an urgent need for multi-center clinical studies with large samples to provide high-quality evidence in the field of prioritizing TIPS for the treatment of acute gastric variceal bleeding.

The present study aims to compare the preemptive TIPS (performed during the first 72 hours after endoscopy) with standard second prophylaxis (endoscopic injection of tissue adhesives plus carvedilol) for patients with acute bleeding from gastric varices (IGV1 or GOV2). The primary outcome will be a 6-week mortality from inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis (diagnosed by imaging, laboratory tests, clinical symptoms, or liver biopsy);
* Admission due to acute bleeding from gastric varices (IGV1 or GOV2).

Exclusion Criteria:

* Prior treatment with TIPS or surgical shunt;
* Presence of contraindications to endoscopic treatment, carvedilol, or TIPS;
* Presence of hepatocellular carcinoma exceeding Milan criteria;
* Presence of other systemic malignant tumors with expected survival time not exceeding 6 months;
* Presence of uncontrollable infection or sepsis;
* Presence of cardiac, pulmonary, or renal failure;
* Pregnant or lactating women;
* Refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6-week mortality | 6 weeks
  The rate of mortality during the first 6 weeks after inclusion in the study.

SECONDARY OUTCOMES:
5-day treatment failure | 5 days
  Incidence of cases requiring adjustment of treatment strategy within 5 days of initial standardised treatment: vomiting of blood or drainage of ≥100 ml of fresh blood from a gastric tube after 2 hours of treatment, hypovolemic shock, drop in haemoglobin of 30 g/L or more within 24 hours without transfusion.
1-year mortality | 1 year
  The rate of mortality during the first 1 year after inclusion in the study.
decompensation events | 1 year
  Rates with rebleeding, new overt ascites (moderate-heavy) or increased degree of ascites, overt hepatic encephalopathy (West-Heaven grades 2-4), or jaundice (total bilirubin >51 mmol/L) from 5 days after initial standardised treatment up to 1 year.
adverse events | 1 year
  Events of various complications such as infections, new tumours, organ failure, peptic ulcers, etc., occurring after randomisation up to the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng Luo, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Escorsell A, Garcia-Pagan JC, Alvarado-Tapia E, Aracil C, Masnou H, Villanueva C, Bosch J. Pre-emptive TIPS for the treatment of bleeding from gastric fundal varices: Results of a randomised controlled trial. JHEP Rep. 2023 Mar 1;5(6):100717. doi: 10.1016/j.jhepr.2023.100717. eCollection 2023 Jun. PMID 37284139